CLINICAL TRIAL: NCT00661245
Title: Transoral Gastroplasty for the Treatment of Morbid Obesity
Acronym: TOGA®
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Satiety, Inc. (Industry)
Responsible Party: Allan L. Abati, Ph.D., VP of RA, QA & Clinical Programs, Satiety, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S107
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TOGA (Experimental): The TOGA procedure is an incision-free treatment using a set of flexible staplers introduced into the mouth and esophagus to create a sleeve in the stomach (transoral formation of a gastric sleeve). The TOGA sleeve limits the amount of food that can be eaten and gives the patient a feeling of fullness after a small meal.
  Interventions: Device: TOGA
- Control (Sham Comparator): A gastric sleeve is not formed.
  Interventions: Device: Control

INTERVENTIONS:
Device: TOGA — Transoral Gastroplasty (TOGA®) System for gastric stapling.
  Arms: TOGA
Device: Control — The control device (bougie dilator) is a FDA-cleared (Class II) device.
  Arms: Control

SUMMARY:
The TOGA® trial is a prospective, multi-center, randomized sham-controlled trial designed to determine the safety and effectiveness of the TOGA System for the treatment of morbid obesity. The study will also determine the effect of the treatment on co-morbidities and quality of life.

Subjects will be blinded to treatment or sham. Sham arm may crossover to TOGA treatment at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60
2. BMI ≥ 40 kg/m2 and < 55 kg/m2, or BMI ≥ 35 kg/m2 with one or more significant co morbidities
3. History of obesity for at least 2.5 years.
4. History of stable weight (defined as a < 10% change in excess weight) for one year prior to the screening visit.
5. History of failure with non-surgical weight loss methods.
6. Suitable candidate for bariatric surgery based on the results of their psychological and physical evaluations.
7. Understands risks of procedure, agrees to follow protocol requirements, including signing informed consent, returning for follow-up visits, completing all required testing, completing diet and behavior modification counseling, committing to prolonged lifestyle changes, and agrees to comply with the substantial dietary restrictions required by the procedure.
8. Subject lives, and intends to remain, within a 100 mile radius of the study center for 5 years.

Exclusion Criteria:

1. Hormonal or genetic cause for the obese state.
2. History of cancer other than localized basal cell carcinoma.
3. History of inflammatory disease of the gastrointestinal tract including Crohn's disease, ulcerative colitis, severe intractable esophagitis, gastric ulceration, or esophageal or duodenal ulceration.
4. Active peptic ulcer disease.
5. Significant known esophageal disease, including Zenker's diverticulum, grade 3-4 reflux esophagitis, stricture, Barrett's esophagus, esophageal cancer, esophageal diverticulum, dysphagia, achalasia, diffuse esophageal spasm, and symptoms of dysmotility.
6. Myocardial infarction or cerebrovascular accident within past year.
7. Angina pectoris.
8. Inability to extend neck or fully open mouth.
9. Clinically severe cervical spinal disease, including cervical disc disease, vertebral osteophytes.
10. Critically loose teeth.
11. Temporomandibular joint syndrome (TMJ) or patients at risk for developing TMJ.
12. Severe coagulopathy (prothrombin time > 3 seconds over control or platelet count < 100,000)
13. Gastroparesis
14. Upper GI bleeding conditions such as esophageal or gastric varices, portal hypertensive gastropathy, congenital or acquired intestinal telangiectasis.
15. Congenital or acquired anomalies of the GI tract such as atresias or stenoses.
16. Structural abnormalities of the GI tract such as diverticulum.
17. Lesions with increased risk of bleeding.
18. Hiatal hernia ≥ 2cm.
19. Severe cardiopulmonary disease or other serious organic disease, including HIV or cancer.
20. Congestive heart failure.
21. Uncontrolled hypertension (systolic >150 or diastolic > 100).
22. Advanced rheumatoid arthritis.
23. Severe or advanced liver disease (such as cirrhosis, chronic hepatitis, portal hypertension, etc.).
24. Chronic pancreatitis.
25. Any contraindication to endoscopy.
26. Severe reflux disease.
27. Currently pregnant or nursing.
28. Potentially childbearing (i.e. not post-menopausal or surgically sterilized) and not willing to use an effective method of contraception for the next 24 months.
29. Alcohol (> 80 gm/day of ethanol) or illicit drug use within the last 3 years.
30. Prior gastric, esophageal, pancreatic or bariatric surgery.
31. Currently on prescription or over the counter diet drugs.
32. Chronic therapy with aspirin, NSAID or anticoagulants.
33. Systemic infection at the time of the procedure.
34. Patient with a known diagnosis or pre-existing symptoms of autoimmune connective tissue disease (i.e., systemic lupus erythematosus or scleroderma).
35. Thyroid disease which is not controlled with medication
36. Unacceptable medical risk (general health status would preclude surgery should a complication occur).
37. Not ambulatory.
38. Participating in another ongoing clinical trial in which concomitant diagnosis or therapeutic intervention would adversely affect the integrity of the clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 275 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Effectiveness: The proportion of subjects with ≥ 25% EWL (excess weight loss); Safety: Pre-defined objective performance criteria (OPC) | 12 months

SECONDARY OUTCOMES:
Improvement in Co-morbidities; Improvements in other Obesity Measures and in Quality of Life Measures | 12 months

CONTACTS AND LOCATIONS:
Locations (11):
- United States (10):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - UMass Memorial Medical Center (University of Massachusetts), Worcester, Massachusetts
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - University of Missouri Health Care, Columbia, Missouri
  - Washington University in St. Louis - School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - University Hospitals Geauga Medical Center, Chardon, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - University of Texas Medical School at Houston, Houston, Texas
- Hospital Erasme, Universite Libre de Bruxelles, Brussels, Belgium